CLINICAL TRIAL: NCT06405191
Title: The Effect of Web-based Education on Psychomotor Skills Education in Nursing; Randomized Controlled Experimental Trial
Brief Title: The Effect of Web-based Education on Psychomotor Skills Education in Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, HAslan [Hakime ASLAN] Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: hakime aslan
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Nursing; Education

STUDY DESIGN:
Intervention Model Description: Randomized cotrolled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web Based Group (Experimental): For 2 weeks, a web-based education intervention was implemented.
  Interventions: Behavioral: Web based education
- Control Group (No Intervention): No intervention was applied to the students in the control group.

INTERVENTIONS:
Behavioral: Web based education — The link to the web page was shared with the students in the experimental group (https://inonuhemsirelikesaslari.com, the expired page cannot be accessed at the moment). Theoretical training and application process steps video for IV catheterization and IM injection skills were taken to the students in the experimental group and uploaded to the web page. The students in the experimental group were given a username-password with which they could access the web page, and the access status of the students was followed by the researcher. The researcher was able to see the frequency of each student watching the videos and their scores in online tests. The student who did not watch the videos or did not take the test was interviewed and feedback was given about watching them. Students were able to access the web page as often as they wanted for two weeks.
  Arms: Web Based Group

SUMMARY:
Objective: This research was conducted to evaluate the effect of web-based education on psychomotor skills teaching and information levels in nursing students.

Materials and Methods: The study was conducted as a randomized controlled clinical trial. The universe of the research consisted of first-year students of the nursing department of a university. The sample of the study consisted of 90 students, experimental and control group. At the beginning of the study, the drug administration course was explained theoretically to all students. Psychomotor skill teaching was demonstrated to both groups in the laboratory with demonstration technique. Then, pre-test data were collected. Students in the experimental group were given a link to the web page where they could watch the clinical knowledge and skills teaching video and a user profile was created. The students had the opportunity to watch and repeat the training videos and lecture notes as much as they wanted for two weeks. In the last stage, the knowledge and skill level of both groups was measured again and post-test data were collected. In order to collect data, intravenous-intramuscular injection skill checklists and drug administration knowledge tests created by the researchers were used.

DETAILED DESCRIPTION:
In today's conditions, depending on the developments in computer and technology, it is inevitable to utilise internet technologies in teaching environments. At this point, Web Based Education (WBE) applications emerged with the use of internet technologies. Many education institutions, especially at higher education level, continue to carry out serious research and development studies in this field as well as realising WBE applications. It was observed that the knowledge level of first-year nursing students about drug applications, intramuscular injection and intravenous catheter insertion skills can be improved with web-based education.

ELIGIBILITY:
Inclusion Criteria:

* Students who volunteered to participate in the research,
* who took the nursing basics course for the first time,
* who did not graduate from a health vocational high school or any associate or undergraduate degree related to health departments,
* who had internet access,
* who had a smart phone or computer were included in the study.

Exclusion Criteria:

* Having any psychological diagnosis,
* İncomplete or incorrect filling of the forms.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Effect of IV catheterization skills | 2 weeks
  IV catheterization; Students in the web-based education group will watch videos, read course materials and solve questions about IV catheterisation practice for 2 weeks.
Effect of IM injection skills | 2 weeks
  IM injection; Students in the web-based education group will watch videos, read course materials and solve questions about IM injection skills for 2 weeks.
Effect of information levels | 2 weeks
  Information levels;Students in the web-based education group will watch videos, read course materials and solve questions about IM injection skills and IV catheterisation practice for 2 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Hakime Aslan, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslan H, Erci B. The effect of playing games with toys made with medical materials in children with cancer on pain during intravenous treatment. Palliat Support Care. 2022 Feb;20(1):84-93. doi: 10.1017/S1478951521000390. PMID 33947501